CLINICAL TRIAL: NCT01298479
Title: Quantitative Determination of the Volume of Suspension Delivered Via the Uniject Delivery System Following Simulated Subcutaneous Injection by Healthcare Professionals Into a Synthetic Subcutaneous Injection Training Device
Brief Title: Sayana-Uniject Volumetric Delivery
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6791034
Record Dates: First submitted 2010-12-16; First posted 2011-02-17 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Volume Delivery
Keywords: volume delivery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: All subjects
  Interventions: Other: Uniject

INTERVENTIONS:
Other: Uniject — single use container

SUMMARY:
The purpose of this study is to determine the volumetric delivery of the Uniject.

DETAILED DESCRIPTION:
Observe subjects deliver the drug None used

ELIGIBILITY:
Inclusion Criteria:

* Nurses

Exclusion Criteria:

* Non-nurses

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: nurses
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Weight of drug suspension delivered (estimated by change in mass of the Uniject(TM) delivery system). | Visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6791034&StudyName=Sayana-Uniject%20Volumetric%20Delivery